CLINICAL TRIAL: NCT03201913
Title: Phase 1 Study of TTC-352 in Patients With Metastatic Breast Cancer Progressing on Endocrine Therapy
Brief Title: Study of TTC-352 in Patients With Metastatic Breast Cancer Progressing on Endocrine Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TTC Oncology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTC-352-101
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Metastatic ER+ Breast Cancer

STUDY DESIGN:
Intervention Model Description: Open-label, accelerated dose escalation study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Accelerated dose escalation study (Experimental): Dose escalation of TTC-352 administered as an oral capsule, twice a day for 28 days (one cycle).
  Patients will receive sequential 28-day cycles of treatment until disease progression, unacceptable toxicity, patient refusal to continue treatment, any other reason to discontinue treatment (e.g., further participation is not in the patient's best interest) or study completion/termination.
  Interventions: Drug: TTC-352

INTERVENTIONS:
Drug: TTC-352 — Phase 1 study to determine the maximum tolerated dose (MTD) of TTC-352.
  Other Names: Selective Human Estrogen Receptor Partial Agonist

SUMMARY:
Phase1 study of TTC 352 for treatment of metastatic ER+ breast cancer.

DETAILED DESCRIPTION:
This is open-label, accelerated dose escalation study of TTC 352, a selective human ER partial agonist for treatment of metastatic ER+ breast cancer in patients who received and progressed on at least two lines of endocrine therapy with one that included a CDK4/CDK6 inhibitor.

The primary objective of this study is to determine the maximum tolerated dose (MTD) of TTC-352 for the treatment of metastatic ER+ breast cancer progressing after endocrine therapy.

The maximum tolerated dose (MTD) of TTC-352 will be determined using initial single-patient cohort escalations until grade 2 toxicity, then expansion to a modified-Fibonacci dose-escalation 3+3 design. Patients enrolled at each dose escalation step must complete the first 28-day cycle of treatment without a dose-limiting toxicity (DLT), or be withdrawn because of a DLT, before additional patients may be enrolled for the next dose escalation step. The MTD dose level cohort will be expanded to a total of 9 patients, to further evaluate safety. In each cohort pharmacokinetics of TTC-352 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. be ≥18 years of age;
2. have a diagnosis of metastatic ER+ breast cancer in patients who received and progressed on at least two lines of endocrine therapy, with one that included a CDK4/CDK6 inhibitor (e.g., palbociclib or ribociclib);
3. have metastatic disease evaluable on imaging studies;
4. have a histologically confirmed diagnosis of ER+ breast cancer;
5. have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1 (Appendix II);
6. have adequate hepatic function, defined as having a serum total bilirubin concentration ≤1.5mg/d, or ≤2 x the upper limit of normal (ULN) if associated with hepatobiliary metastases or Gilbert syndrome, and having serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) concentrations ≤2.5 × ULN, or ≤5 x ULN for patients with known hepatic metastases;
7. have adequate renal function, defined as having a serum creatinine ≤1.5 × ULN and a creatinine clearance ≥40mL/min (estimated using the Cockcroft-Gault formula);
8. have adequate hematologic function, defined as having a hemoglobin ≥8g/dL, an absolute neutrophil count (ANC) ≥1.0 × 109/L, and platelet count ≥75.0 x 109/L;
9. be willing and able to comply with study visits and procedures;
10. have read, understood and signed the informed consent form (ICF) approved by the Institutional Review Board (IRB);
11. if a woman of childbearing potential (WOCP), not be pregnant (confirmed by a negative serum pregnancy test within 14 days of study entry and re-confirmed by a urine pregnancy test on the morning of Study Day 1, prior to the start of study treatment) and/or not be breast-feeding; [Note: Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) are not considered to be a WOCP.]
12. If a WOCP, agree to use during the study and for at least one month after the last dose of study drug a medically acceptable method of birth control [such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence.];
13. if male (and whether or not surgically or medically sterile), agree to use during the study and for at least one month after the last dose of study drug a double barrier method of birth control (in addition to any other birth control method practiced by his partner) while engaging in sexual intercourse with a partner who is pregnant, possibly pregnant or able to become pregnant.

Exclusion Criteria:

1. have received chemotherapy, hormonal therapy, biologic therapy, immunotherapy or radiation therapy within 14 days prior to the planned start of study treatment.
2. have inadequate recovery* from adverse events resulting from previously-administered anti-cancer therapies; [*Note: Unless more specifically defined in Inclusion Criteria 6, 7 and 8 above, adequate recovery is defined as improvement to ≤ Grade 2 for any other hematologic toxicity and for peripheral neuropathy, and improvement to ≤ Grade 1 for any other non-hematologic toxicity.]
3. have a history of venous thromboembolism, including deep vein thrombosis, pulmonary embolism or retinal vein thrombosis, unless currently on anticoagulant therapy;
4. have impending visceral crisis that requires chemotherapy;
5. have known uncontrolled or symptomatic CNS metastases;
6. have any clinically significant infection, defined as any acute viral, bacterial, or fungal infection that requires systemic treatment or have received any anti-infective treatment within 7 days prior to the screening visit;
7. have any other severe, uncontrolled medical condition, including unstable congestive heart failure (Stage III-IV of the New York Heart Association Functional Classification (Appendix III))
8. have a known or suspected allergy to the study drug or any study drug component;
9. have any other medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, that may interfere with the interpretation of study results or that otherwise would, in the opinion of the Investigator, make study participation inappropriate;
10. have any non-healing wound, fracture, or ulcer within 28 days prior to the planned start of study treatment;
11. have received any other investigational drug within 28 days (or 5 half-lives, if longer) prior to the start of study screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
MTD | 24 months
  The primary objective of this study is to determine the maximum tolerated dose (MTD) of TTC-352 for the treatment of metastatic ER+ breast cancer progressing after endocrine therapy

SECONDARY OUTCOMES:
Best response to treatment | 24 months
  Determine patient best response to treatment (complete response, partial response, stable disease or disease progression) after at least two 28-day cycles of treatment with TTC 352.
PFS | 24 months
  Determine durations of progression-free survival after at least two 28-day cycles of treatment with TTC 352
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
  Treatment-related adverse events as assessed by CTCAE v4.0 will be collected in presented in tabular form at the end of study.
Maximum Plasma Concentration (Cmax) | 24 months
  Blood samples will be collected at the following Cycle 1 time points:
  Day 1: prior to dosing and at Hours 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 after dosing (just before dosing on Day 2).
  Day 28: prior to dosing and at Hours 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 28 after dosing.
  TTC-352 blood levels will be measured at above time points and Cmax will be calculated.
Half life | 24 months
  Blood samples will be collected at the following Cycle 1 time points:
  Day 1: prior to dosing and at Hours 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 after dosing (just before dosing on Day 2).
  Day 28: prior to dosing and at Hours 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 28 after dosing.
  TTC-352 blood levels will be measured at above time points and half life of TTC-352 will be calculated.
Area Under the Curve (AUC) | 24 months
  Blood samples will be collected at the following Cycle 1 time points:
  Day 1: prior to dosing and at Hours 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 after dosing (just before dosing on Day 2).
  Day 28: prior to dosing and at Hours 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 28 after dosing.
  TTC-352 blood levels will be measured at above time points and AUC will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Z Dudek, MD, Study Chair — TTC Oncology, LLC
Locations (4):
- United States (4):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - HealthPartners Institute, Regions Cancer Care Center, Saint Paul, Minnesota
  - Sanford Health, Sioux Falls, South Dakota
  - University of Wisconsin, Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
At present TTC Oncology does not plan to share IPD with other researchers.

REFERENCES:
- [Derived] Dudek AZ, Liu LC, Fischer JH, Wiley EL, Sachdev JC, Bleeker J, Hurley RW, Tonetti DA, Thatcher GRJ, Venuti RP, O'Regan RM. Phase 1 study of TTC-352 in patients with metastatic breast cancer progressing on endocrine and CDK4/6 inhibitor therapy. Breast Cancer Res Treat. 2020 Oct;183(3):617-627. doi: 10.1007/s10549-020-05787-z. Epub 2020 Jul 22. PMID 32696319